CLINICAL TRIAL: NCT01120496
Title: A Randomized Controlled Trial of Nebulized Hypertonic Saline Treatment in Hospitalized Children With Moderate to Severe Viral Bronchiolitis
Brief Title: Nebulized Hypertonic Saline Treatment in Hospitalized Children With Moderate to Severe Viral Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: zhengxiu luo, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChiCTR-TRC
Record Dates: First submitted 2010-04-23; First posted 2010-05-11 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2008-11

CONDITIONS: Bronchiolitis
Keywords: Hypertonic saline solution, bronchiolitis, RSV
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypertonic saline (Experimental): hypertonic saline (HS)
  Interventions: Drug: 3% hypertonic saline
- normal saline (NS) (Placebo Comparator): normal saline (NS)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: 3% hypertonic saline — Moderately to severely ill infants with bronchiolitis were randomized to receive 4 mL solution containing either 3% hypertonic saline or normal saline
  Other Names: normal saline
  Arms: hypertonic saline
Drug: normal saline — Moderately to severely ill infants with bronchiolitis were randomized to receive 4 mL solution containing either 3% hypertonic saline or normal saline
  Other Names: 3% hypertonic saline
  Arms: normal saline (NS)

SUMMARY:
The purpose of this study is planned to investigate whether frequently inhaled hypertonic saline (HS) can relieve symptoms and signs faster than normal saline (NS) and shorten length of stay (LOS) significantly for moderately to severely ill infants with bronchiolitis without apparent adverse effects.

DETAILED DESCRIPTION:
The treatment of bronchiolitis remains largely supportive with mechanical ventilatory support as needed .Other types of treatment remain controversial.We and other researchers have demonstrated that nebulized HS and bronchodilators decreased symptoms and LOS for infants with mild to moderate viral bronchiolitis .All the aforementioned studies used 3 times per day dosing, which is significantly less than the 3 to 6 times per hour regimens often used in children in respiratory distress.Frequently nebulized HS reduced the LOS for infants with moderately severe bronchiolitis.The present study is planned to investigate whether frequently inhaled HS can relieve symptoms and signs faster than NS and shorten LOS significantly for moderately to severely ill infants with bronchiolitis without apparent adverse effects.

PMID: 15266547 PMID: 12576370 PMID: 16599051 PMID: 17719935 PMID: 20014350 PMID: 12475841

ELIGIBILITY:
Inclusion Criteria:

* infants less than 24 months of age with first episode of wheezing.

Exclusion Criteria:

* age>24 months,
* previous episode of wheezing,
* chronic cardiac and pulmonary disease,
* immunodeficiency,
* accompanying respiratory failure,
* requiring mechanical ventilation,
* inhaling the nebulized 3% hypertonic saline solution 12 hours before treatment,
* premature infants born at less than 34 weeks gestation.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of frequently nebulized HS in moderately to severely ill infants with bronchiolitis | 1 year
  Compare the wheezing remission time,Cough remission time,moist crackles disappeared time and the hospital length of stay between HS and NS.

SECONDARY OUTCOMES:
To determine the safety of frequently nebulized HS in moderately to severely ill infants with bronchiolitis | 1 year
  evaluated for the hoarse voice, vomiting, diarrhea, general condition

CONTACTS AND LOCATIONS:
Overall Officials: zhengxiu luo, doctor, Principal Investigator — Chongqing Medical University

REFERENCES:
- See also: Related Info — http://www.clinicaltrials.gov